CLINICAL TRIAL: NCT00744146
Title: Phase I, Randomized, Controlled, Third-party Double-blind, Dose Escalating Study of Protexia Administered Intramuscularly at One or Two Time Points in Healthy Human Volunteers
Brief Title: First Time in Human Study of Protexia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmAthene, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency); Quintiles, Inc. (Industry); QPS Holdings LLC (Industry)
Responsible Party: Valerie Riddle, M.D., Vice President and Medical Director, PharmAthene, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: QOPK 4439
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2010-09

CONDITIONS: Intervention for Nerve Agent Exposure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): Six volunteers total.
  Randomized such that four volunteers will receive Protexia as a single 50 mg dose and two volunteers will receive saline placebo of the same volume on Study Day 1.
  Volunteers to be followed for approximately 71 days total.
  Interventions: Biological: Protexia
- 2 (Experimental): Six volunteers total.
  Randomized such that four volunteers will receive Protexia as a single 100 mg dose and two volunteers will receive saline placebo of the same volume on Study Day 1.
  Volunteers to be followed for approximately 71 days total.
  Interventions: Biological: Protexia
- 3 (Experimental): Eight volunteers total.
  Randomized such that six volunteers will receive Protexia as a single 250 mg dose and two volunteers will receive saline placebo of the same volume on Study Days 1 and 72.
  Volunteers to be followed for approximately 142 days total.
  Interventions: Biological: Protexia
- 4 (Experimental): Six volunteers total.
  Randomized such that four volunteers will receive Protexia as a single 500 mg dose and two volunteers will receive saline placebo of the same volume on Study Day 1.
  Volunteers to be followed for approximately 71 days total.
  Interventions: Biological: Protexia
- 5 (Experimental): Six volunteers total.
  Randomized such that four volunteers will receive Protexia as a single 750 mg dose and two volunteers will receive saline placebo of the same volume on Study Day 1.
  Volunteers to be followed for approximately 71 days total.
  Interventions: Biological: Protexia

INTERVENTIONS:
Biological: Protexia — Single 50 mg IM dose
  Other Names: PEG-rBChE
  Arms: 1
Biological: Protexia — Single 100 mg dose
  Other Names: PEG-rBChE
  Arms: 2
Biological: Protexia — Two 250 mg doses, IM, one at Day 1 and one at Day 72
  Other Names: PEG-rBChE
  Arms: 3
Biological: Protexia — Single 500 mg dose, IM
  Other Names: PEG-rBChE
  Arms: 4
Biological: Protexia — Single 750 mg dose, IM
  Other Names: PEG-rBChE
  Arms: 5

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and immunogenicity of Protexia, an experimental drug being developed to protect soldiers against the effects of nerve agents.

Volunteers will be entered into one of five groups. Four of the groups will receive a single intramuscular dose of Protexia or saline placebo on Study Day 1 and will participate in the study for approximately 71 days. One of the groups will receive two intramuscular doses of Protexia or saline placebo - one dose on Study Day 1 and the second dose on Study Day 72. This group will participate in the study for approximately 142 days.

All volunteers will remain at the study site as an inpatient for three days after they are dosed and will be monitored closely by the study doctors and staff. After that, volunteers will return to the study site as outpatients at predetermined intervals. Groups 1, 2, 4, 5 will have a total of 6 follow-up visits and Group 3 will have a total of 12 follow-up visits.

It is expected that this study will provide important information on the safety and tolerabiity of Protexia at one and two doses.

DETAILED DESCRIPTION:
Protexia is a pegylated form of recombinant human butyrylcholinesterase (PEG-rBChE). Butyrylcholinesterase (BChE) is a naturally-occurring enzyme found in minute quantities in the blood. PharmAthene produces PEG-rBChE from the milk of transgenic goats. The enzyme is purified from the goat milk, formulated and pegylated to create Protexia.

This is a dose escalation study of five dose levels of Protexia. Safety data through 14 days post-dosing will be evaluated by an independent Safety Monitoring Committee (SMC) prior to escalating to a higher dose. The safety and tolerability of Protexia will be assessed using the DMID Adult Toxicity Table, May 2001 (Appendix D).

If a dose limiting toxicity (DLT) is identified in any dosing group, dosing will be suspended until the AE(s) is/are assessed. The SMC will determine if the study can continue or if the previous dose will be declared the maximum tolerated dose (MTD). It is possible that an additional dosing group at a dose midway between the previous dosing group and the dose level that exceeded the MTD may be enrolled after consultation and agreement of the SMC.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers aged 18 to 55 years
* Willing to give written informed consent to participate in the study and to comply with all study requirements and procedures
* In the opinion of the Investigator, in generally good health, based upon pre-study medical history, physical examination, electrocardiogram (ECG) and laboratory tests
* Normal clinical chemistry, hematology and urinalysis results or clinically insignificant values during screening evaluations
* Women of childbearing potential may be enrolled if one of the following criteria applies:

  * Using effective contraception (e.g., injectable, transdermal, vaginal ring, oral contraceptives, IUD or barrier methods) for at least three months prior to study entry, must have maintained a normal menstrual pattern for the 3 months prior to study entry and agree to continue contraception for the duration of their participation in the study.
  * Females using injectable, transdermal, vaginal ring, oral contraceptives or an IUD must agree to augment this with a barrier method for the duration of their participation in the study.
  * Is sexually abstinent
  * Is monogamous with a vasectomized partner
  * Is postmenopausal (i.e., no cycle for at least the previous 24 months and is of menopausal age (> 45 years)
  * Has not had a menstrual cycle for 12 to 24 months and is of menopausal age as described above
  * Is surgically sterilized
  * Has had a total hysterectomy a minimum of 3 months prior to dosing on Day 1
* Females with a negative urine pregnancy test at study Screening and a negative serum pregnancy test on admission to the Phase I unit at Day -1

  * Females in Group 3 will also require a negative serum pregnancy test on Day 71 prior to receiving Dose 2
* Sexually active male subjects may be enrolled if one of the following criteria applies:

  * Has had a vasectomy
  * Using condoms and whose partner is using an acceptable form of contraception (IUD, oral contraceptives, birth control patch or vaginal ring, injectable or implanted contraceptives, or tubal ligation [surgical sterilization]) for the duration of the study
  * Is sexually abstinent
* Body Mass Index (BMI) 19 to 29, inclusive
* Abstinence from alcohol for 24 hours prior to study drug administration until discharge from the Phase I unit on Day 4

Exclusion Criteria:

* Inability to provide Informed Consent
* Drug or alcohol abuse requiring treatment within 12 months of study screening
* Positive drug result at time of study screening or positive alcohol result at Day -1 (and Day 71 for Group 3 subjects)
* Use of cholinesterase inhibitors within 21 days of dosing
* Receipt of fresh frozen plasma within three months of study screening
* Allergy to milk or milk derived products
* History of allergic reaction to procainamide or to its metabolite, p-aminobenzoic acid
* Diagnosis of myasthenia gravis
* Participation in any trial of an investigational agent within 30 days of study screening
* Previous receipt of any investigational BChE product
* Clinically significant medical or psychiatric condition that, in the opinion of the Investigator, may impair study participation
* ECG with evidence of clinically significant conduction abnormalities or active ischemia at time of study screening
* Donation of one or more pints of blood within 30 days prior to study screening
* Known serum positivity for human immunodeficiency virus (HIV) antibodies, hepatitis B or hepatitis C
* Extensive tattooing which would preclude adequate assessment at the injection site(s)
* Females who are pregnant and/or breast feeding
* Use of systemic immunosuppressive agents, such as used to treat Alzheimer's Disease, within 3 months of dosing
* Use of dietary or herbal supplements within 3 months of dosing

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Safety will be assessed by: - The determination of dose limiting toxicity (if reached) - Changes from baseline for clinical laboratory tests, urine tests and vital signs - Descriptive statistics for adverse events and safety parameters | Volunteers in 4 of 5 Groups will be followed for 72 days. Volunteeers in 1 group will be followed for 142 days.

SECONDARY OUTCOMES:
Pharmacokinetics and immunogenicity will be assessed. | Volunteers in 4 of 5 Groups will be followed for 72 days. Volunteeers in 1 group will be followed for 142 days.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph A Schutz, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Quinitles Phase I Services, Overland Park, Kansas, United States